CLINICAL TRIAL: NCT03768713
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Determine the Effect of Suvorexant (Belsomra®) on Sympathetic Neural Activity and Baroreflex Function in Patients With Chronic Insomnia
Brief Title: Impact of Suvorexant on Sympathetic Nerve Activity and Baroreflex Function in Chronic Insomnia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Montana State University (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: JC101320-FC
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug (Suvorexant) (Experimental): 20 mg of Suvorexant daily (taken orally ~1 hour before bedtime)
  Interventions: Drug: Suvorexant
- Placebo (Placebo Comparator): 20 mg of Placebo daily (taken orally ~1 hour before bedtime)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — Insomnia subjects will take a nightly pill of 20 mg Suvorexant for eight weeks.
  Arms: Drug (Suvorexant)
Drug: Placebo — Insomnia subjects will take a nightly pill of 20 mg placebo for eight weeks.
  Arms: Placebo

SUMMARY:
This study aims to evaluate the effect of Suvorexant on sympathetic nerve activity and baroreflex function in subject with chronic insomnia. The investigator's central hypothesis is that Suvorexant will reduce sympathetic nerve activity and improve baroreflex function when compared to placebo.

DETAILED DESCRIPTION:
This study will utilize a randomized, double-blind, placebo-controlled experimental approach to determine the effects of 8-wk treatment with Suvorexant (Belsomra®) on sympathetic nerve activity and baroreflex function in male and female subjects with chronic insomnia. The study will utilize established techniques for assessing sleep (polysomnography), blood pressure (sphygmomanometer and beat-to-beat finger plethysmography), and peripheral sympathetic nerve activity (microneurography). The study will stratify enrollment based upon both age and sex (i.e., male vs. female) because these two covariates are known to influence sympathetic nerve activity and baroreflex function.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 3 months of clinically diagnosed insomnia
* Body mass index ≤35 kg/m2
* Insomnia Severity Index (ISI) > 7 arbitrary units (i.e., mild-to-severe insomnia)
* Pre-menopausal women must have regular menstrual cycles (~26-30 day cycles) and will be scheduled for microneurography 2-7 days after menstruation to consistently test during the early follicular phase (or low-hormone phase in women on contraceptives)

Exclusion Criteria:

* Current or prior treatment of Suvorexant.
* Obstructive sleep apnea defined as an apnea-hypopnea index > 30 using an FDA approved home sleep apnea screening devices as used in routine clinical practice.
* Participants without evidence of clinically significant obstructive sleep apnea on the screening test will undergo an overnight in-laboratory polysomnography to confirm absence of sleep apnea (apnea-hypopnea index of ≥ 30 episodes per hour) and to exclude other sleep disorders (e.g. periodic limb movement arousal index of ≥ 5 episodes per hour)
* Circadian rhythm sleep disorders
* History of meeting DSM-V criteria of major psychiatric disorder
* Have been clinically-diagnosed with diabetes, cardiovascular disease, or any other unstable or serious medical condition.
* Current, or use within past month, of psychoactive (other than stable treatment with antidepressant or antianxiety), hypnotic, stimulant or analgesic medication (except occasional non-narcotic analgesics)
* Shift work or other types of self-imposed irregular sleep schedules
* Habitual smoking (6 or more cigarettes per week)
* Habitual alcohol consumption (more than 2 alcoholic drinks per day)
* Breastfeeding or pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-04-18 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Sympathetic nerve activity | 8 weeks
  Direct recordings of muscle sympathetic nerve activity from the peroneal nerve using a microelectrode.
Baroreflex sensitivity | 8 weeks
  The linear relationship between changes in beat-to-beat diastolic arterial pressure and changes in sympathetic nerve activity.

SECONDARY OUTCOMES:
Sympathetic reactivity | 8 weeks
  The change in muscle sympathetic nerve activity during a cold pressor test.
Home sleep quality: Wrist actigraphy | 8 weeks
  Wrist actigraphy will be used to to determine the quality of sleep, with a primary focus on sleep efficiency.
Laboratory sleep quality: Polysomnography | 8 week
  Polysomnography will be used to determine the quality of sleep, with a primary focus on sleep efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Carter, PhD, Principal Investigator — Montana State University
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No